CLINICAL TRIAL: NCT07099430
Title: An Open-label, Multicenter Phase Ib/II Clinical Study to Evaluate the Efficacy and Safety of LBL-024 Monotherapy, LBL-024 in Combination With LBL-007 or Toripalimab in Patients With Advanced Melanoma
Brief Title: A Trial of LBL-024 Monotherapy, LBL-024 Combined With LBL-007 or Toripalimab in Patients With Advanced Melanoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Leads Biolabs Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LBL-024-CN007
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-09

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Injections; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LBL-024 (Experimental): Cohort 1 (LBL-024 monotherapy):
  Subjects received treatment with LBL-024 , intravenous infusion.
  Interventions: Drug: LBL-024 for Injection
- LBL-024 + LBL-007 combination (Experimental): Cohort 2 (LBL-024 + LBL-007 combination):
  Subjects received treatment with LBL-024 combined with LBL-007 , intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: LBL-007 Injection
- LBL-024 + toripalimab combination (Experimental): Cohort 3 (LBL-024 + toripalimab combination ):
  Subjects received treatment with LBL-024 combined with toripalimab , both intravenous infusion.
  Interventions: Drug: LBL-024 for Injection; Drug: Toripalimab Injection

INTERVENTIONS:
Drug: LBL-024 for Injection — LBL-024 , Intravenous infusion.
  Other Names: LBL-024
Drug: LBL-007 Injection — LBL-007 , intravenous infusion.
  Other Names: LBL-007
  Arms: LBL-024 + LBL-007 combination
Drug: Toripalimab Injection — Toripalimab , intravenous infusion.
  Other Names: Toripalimab
  Arms: LBL-024 + toripalimab combination

SUMMARY:
This study is an open-label, multicenter phase Ib/II study to evaluate the efficacy and safety of LBL-024 monotherapy, LBL-024 in combination with LBL-007 or toripalimab in patients with advanced melanoma,To evaluate the preliminary efficacy and safety of LBL-024 monotherapy and combination therapy in patients with advanced melanoma.

DETAILED DESCRIPTION:
This trial includes two phases, Phase Ib and Phase II.

Phase Ib is an exploratory stage of safety and efficacy in a single-arm, open-label study, including three cohorts (different dosing regimens).Phase Ib includes three cohorts, Cohort 1 (LBL-024 monotherapy), Cohort 2 (LBL-024 + LBL-007 combination) and Cohort 3 (LBL-024 + toripalimab combination).

Phase II includes Part A and Part B.Part A is a randomized, open-label, positive-controlled extension study. It plans to enroll patients with melanoma of the cutaneous, Acral, and unknown primary. Eligible subjects will be randomly assigned in a 2:1 ratio [Stratification factor: Acral subtype (Yes vs. No)] to either the Experimental Group or the Control Group. Part B is a single-arm extension study enrolling only patients with mucosal melanoma,and will select a drug combination based on phase Ib efficacy for expansion study.

This study requires subjects to provide relevant samples for testing. The trial will enroll up to 200 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to follow the trial treatment regimen, visit schedule,laboratory test, and comply with other requirements of the protocol, and voluntarily enroll in the study and sign the written informed consent.
2. At the time of signing the informed consent form, the age was ≥ 18 years old, and the gender was not limited.
3. The Eastern Cooperative Oncology Group's physical status scoring standard (ECOG) is 0~1.
4. The expected survival time is at least 12 weeks.
5. According to the evaluation of RECIST 1.1 （Response Evaluation Criteria in Solid Tumours）, the subjects enrolled have at least one measurable neoplasm lesion.
6. Male of childbearing potential and Females of childbearing age are willing to take highly effective contraceptive measures From the signing of the informed consent form to within 6 months after the last administration of the trial drug.

Exclusion Criteria:

1. Subjects who received live vaccination within 4 weeks before the first dose or were planned to receive live vaccination during the study period and 4 weeks after the dose.
2. Major surgery or other treatment or diagnosis that has a significant impact on the subject within 4 weeks before the first dose.
3. Patients with active, or who have had and have the possibility of recurrence of autoimmune diseases.
4. History of severe cardiovascular and cerebrovascular disorder.
5. Active infectious disease.
6. History of mental illness (interfering with understanding or giving informed consent), drug abuse, alcoholism, or drug addiction.
7. Women during pregnancy or lactation.
8. The investigator believes that the subject has other conditions that may affect compliance or are not suitable for participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse event (AE) and serious adverse event (SAE) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (90 days after drug withdrawal or before the start of new anti-tumor therapy)
  Adverse event (AE) will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 5.0.The safety profile of LBL-024 monotherapy or combination therapy will be assessed by monitoring the adverse event (AE) and serious adverse event (SAE) in Phase Ib study.
Objective Response Rate (ORR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour) ,Proportion of subjects achieving complete response (CR) or partial response (PR).It was used to evaluate the efficacy in Phase Ib.
Progression-free Survival(PFS) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  According to the evaluation criteria of RECIST V1.1 (solid tumour),Time from first dose to disease progression or death from any cause.It was used to evaluate Time of disease no-progression or Drug resistance in Phase II.

SECONDARY OUTCOMES:
Cmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Maximum drug concentration in plasma after administration.
Tmax | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  After administration,Time to reach maximum drug concentration in plasma.
Immunogenicity | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  The immunogenicity is evaluated by the incidence of anti-drug antibodies (ADA) and neutralizing antibodies (if applicable) in subjects.Immunogenicity refers to the performance that can elicit an immune response.
Disease Control Rate(DCR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  Percentage of participants achieving CR, PR, iCR, iPR and stable disease (SD) after treatment.
Duration of Response(DOR) | From all subjects signed the informed consent form up to the completion of the follow-up period of drug withdrawal (28 days after drug withdrawal or before the start of new anti-tumor therapy)
  DOR is defined as the duration from earliest date of disease response (CR、PR 、iCR or iPR) until earliest date of disease progression or death from any cause(if occurring sooner than progression).

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chen, Principal Investigator — Fujian Cancer Hospital
Locations (15):
- China (15):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute &Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No